CLINICAL TRIAL: NCT05101460
Title: An All Comers Registry For Normothermic Ex Vivo Lung Perfusion (EVLP) as Assessment of Donor Lungs for Transplant
Status: Recruiting | Type: Observational
Sponsor: XVIVO Perfusion (Industry)
Responsible Party: Sponsor
Other Study IDs: XVO-003
Record Dates: First submitted 2021-10-05; First posted 2021-11-01 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-06

CONDITIONS: Lung Transplant
Keywords: Lung Transplant; Transplantation lung
MeSH Terms: interventions — Photoelectron Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: XVIVO Perfusion System (XPS™) with STEEN Solution™ — XVIVO Perfusion System (XPS™) with STEEN Solution™

SUMMARY:
The XVIVO Registry is to collect standard of care clinical data from "all-comers" who are transplanted with an EVLP lung treated with the XVIVO Perfusion System™ in order to assess the long-term performance of the device, and monitor device-related serious adverse events. In addition, 4 and 5-year UNOS registry data of the 126 subjects who received an EVLP transplant under the NOVEL and NOVEL Extension studies are provided as part of the long-term safety and quality of life data. In addition, 4 and 5-year UNOS registry data of the 126 subjects who received an EVLP transplant under the NOVEL and NOVEL Extension studies are provided as part of the long-term safety and quality of life data.

DETAILED DESCRIPTION:
The XVIVO registry is an ongoing, observational, multicenter, retrospective review of patients exposed to XPS™ EVLP-treated lungs. The Registry study is aligned and managed by the UNOS and OPTN data collection process. This registry uses quarterly STAR file data requests for the OPTN data managed by UNOS.

The EVLP procedure and transplantation will be performed per XPS™ Instructions for Use and the treating physician's discretion. Post-transplant clinical care will follow the institution's standard-of-care policies.

OPTN updated the data collected since the submission of the protocol therefore the data collection has changed. The following data has updated collection:

* Collects if hospitalized since last follow-up (yes, no), not the number of hospitalizations
* Collects acute rejection episodes (yes treated, yes not treated, no), not the number of episodes
* Collects Karnofsky Score as replacement for Physical and functional capacity
* Employment limitations has been updated to working for income (yes or no)
* No longer collects BOS, XVIVO to request BOS evaluations on subjects with visits prior to June 30, 2020 and any other omissions of end points not available in the data requested via STAR request.
* Collects FEV1 (L) effective June 30, 2020 to calculate CLAD and diagnosis of CLAD, if applicable.
* No longer provides Other, Specify text in STAR request.

ELIGIBILITY:
This is an "All Comers Registry" hence will include all patients receiving EVLP lungs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an "All Comers Registry" hence, no specific investigator sites. All patients receiving EVLP lungs treated with XPS™ will be included in the registry without eligibility criteria or pre-selection. Since the registry collects only standard-of-care data and requires no additional procedures or risks to the subject, a waiver of consent is appropriate
Sampling Method: Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2019-10-29 (Actual); Primary Completion 2024-04-24 (Estimated); Study Completion 2029-04-24 (Estimated)

PRIMARY OUTCOMES:
Survival at 1 year post-transplant | 12 months
  Primary effectiveness endpoint
Primary Graft Dysfunction (PGD) | 72 hours
  Rate of Grade 3 Primary Graft Dysfunction (PGD) at 72 hours

SECONDARY OUTCOMES:
Post-transplant survival | 2 years, 3 years, 4 years and 5 years post-transplant
  Survival at 2, 3, 4 and 5 years post-transplant
Pulmonary Function Test (FEV1) | 1 year, 2 years, 3 years, 4 years and 5 years post-transplant
  Pulmonary Function Test (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEV1 is the key lung function test in diagnosing BOS. FEV1 test at 1 year, 2 years, 3 years, 4 years and 5 years post-transplant.
Incidence of Bronchiolitis Obliterans Syndrome (BOS) or Chronic Lung Allograft Dysfunction (CLAD) | 1 year, 2 years, 3 years, 4 years and 5 years post-transplant
  Rate of Grade 0 through 3 Bronchiolitis Obliterans Syndrome (BOS) at 1 year, 2 years, 3 years, 4 years and 5 years post-transplant. Clinically, BOS is associated with a progressive decline in forced expiratory volume in one second (FEV1) greater than or equal to 20% of baseline. Decline in FEV1 % increases the risk of development of BOS (Grade 0 to 3).
  CLAD is defined as a substantial and persistent decline (≥ 20%) in measured FEV1 value from the reference (baseline) value after lung transplantation, with or without a change in FVC. If CLAD is identified, staging and phenotype will be assigned.
Hospitalizations | 1 year, 2 years, 3 years, 4 years and 5 years post-transplant
  The presence of in-patient hospital admissions between transplant and 1 year, 1-2 years, 2-3 years, 3-4 years, and 4-5 years post-transplant
Acute Rejection Episodes | 1 year, 1-2 years, 2-3 years, 3-4 years, and 4-5 years post-transplant
  The presence of biopsy proven hospital admissions between transplant and 1 year, 1-2 years, 2-3 years, 3-4 years, and 4-5 years post-transplant
Karnofsky Performance Status Scale (KPS)/Karnofsky score | 1 year, 2 years, 3 years, 4 years and 5 years post-transplant
  Karnofsky Performance Status Scale is an assessment tool for functional impairment. It is used to improve understanding of patient needs, ability to carry out daily activities and to assess patient prognosis. Karnofsky score is calculated at 1 year, 2 years, 3 years, 4 years and 5 years post-transplant. Higher the Karnofsky score, better the ability to carry out daily activities.
Safety Endpoint | 30 days post-transplant
  XPS related SAEs from transplant to 30 days post-transplant or initial hospital stay, whichever is longer

CONTACTS AND LOCATIONS:
Overall Officials: Jaya Tiwari, BS, CCRP, Study Director — XVIVO Perfusion Inc.
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No